CLINICAL TRIAL: NCT03998475
Title: Implementing a Transition Preparation Intervention for Young Adults With Type 1 Diabetes in an Integrated Healthcare Setting
Brief Title: Transition Preparation Intervention for Young Adults With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Commonwealth University (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: HM20015399; 1-19-PDF-041-R (Other Grant/Funding Number: American Diabetes Association)
Record Dates: First submitted 2019-06-24; First posted 2019-06-26 (Actual); Last update posted 2020-11-09 (Actual); Status verified 2020-11

CONDITIONS: Type 1 Diabetes
Keywords: Transition; Young Adult
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Transition preparation program (Experimental): Transition preparation intervention for young adults with type 1 diabetes (T1D)
  Interventions: Behavioral: Transition preparation intervention

INTERVENTIONS:
Behavioral: Transition preparation intervention — Young adult participants and parents will complete transition preparation sessions that include meeting with a health behavior coach for in-person sessions and review of materials sent electronically between study visits.

SUMMARY:
The purpose of this research study is to find out more about how to support young adults (ages 18-22) with type 1 diabetes as they prepare to transition from pediatric and adult endocrinology medical care.

DETAILED DESCRIPTION:
The overarching goal of the proposed trial is to improve diabetes self-management and glycemic control in young adults and prepare them for the transition to adult endocrinology. The current application will investigate the impact of a multisystem transition preparation intervention for young adults (ages 18-22) with T1D. Twenty-five young adults and a parent will be enrolled in a 6-month transition preparation program which will use a hybrid in-person and technology delivery structure. Providers will receive training highlighting their role preparing young adults for transition and provides practical tips to use in their communication with young adults. If effective, this multisystem intervention, designed to enhance T1D self-management and increase young adults' readiness for transition to adult healthcare during this critical developmental period, has the potential to inform clinical practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

Both members of the youth/parent dyad must meet all eligibility criteria

Young adults

* English-speaking
* patients in Pediatric Endocrinology at Children's Hospital of Richmond (CHoR) at Virginia Commonwealth University (VCU)
* between ages 18-22 yrs with a
* diagnosis of T1D for >1 year

Parents

* greater than 18 years of age
* provide care to the young adult with T1D
* are willing to participate in the intervention

Medical providers

• provide care to patients with T1D ages 18-22 yrs in Pediatric Endocrinology at CHoR

Exclusion Criteria:

Young adults

* significant psychiatric, cognitive, medical or developmental conditions that would impair their ability to complete assessments and/or engage in diabetes self-care behaviors (e.g., malignancies, psychosis, intellectual disability), as documented in the medical record or revealed during eligibility screening, or
* medically-induced diabetes or diagnosis of diabetes other than type 1 diabetes

Parents

* non-English speaking
* psychiatric, cognitive, or developmental conditions that would impair their ability to complete assessments and/or engage in the intervention as determined at study screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2019-07-11 (Actual); Primary Completion 2020-09-16 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Number of sessions attended | 6 months
  Number of study visits (attendance)
Number of session views | 6 months
  Number of opened electronic materials (e.g., opened messages in the patient health portal))
Program acceptability - young adult | 9 months
  Young adult report on satisfaction with the program via an exit survey
Program acceptability - parent | 9 months
  Parent report on satisfaction with the program via an exit survey
Program acceptability - provider | 9 months
  Provider report on satisfaction with the program via an exit survey

SECONDARY OUTCOMES:
Change in Glycemic control | Baseline to 9 months
  Measurement of hemoglobin A1c (A1c; reported as a percentage)
Diabetes-related hospitalizations | 9 months
  Participant report and medical record review of count of reported diabetes-related hospitalizations and complications
Change in adherence to diabetes care regimen | Baseline to 9 months
  Average of young adult and parent participant reports on the Diabetes Management Questionnaire (DMQ)
Change in transition readiness | Baseline to 9 months
  Average of young adult and parent participant reports on the Transition Readiness Assessment Questionnaire (TRAQ)

OTHER OUTCOMES:
Change in diabetes self-efficacy | Baseline to 9 months
  Participant (young adult) report on the Self-Efficacy for Diabetes Self-Management (SEDSM)
Change in diabetes quality of life | Baseline to 9 months
  Participant (young adult) report on the Pediatric Quality of Life Diabetes Module
Change in diabetes family responsibility | Baseline to 9 months
  Average of young adult and parent participant reports on the Diabetes Family Responsibility Questionnaire (DFRQ)
Change in diabetes family conflict | Baseline to 9 months
  Average of young adult and parent participant reports on the Diabetes Family Conflict Scale (DFCS)
Change in depression | Baseline to 9 months
  Participant (young adult) report on the Center for Epidemiologic Studies Depression Scale (CESD)
Change in young adult diabetes distress | Baseline to 9 months
  Participant (young adult) report on the Diabetes Distress Scale
Change in parent diabetes distress | Baseline to 9 months
  Participant (parent) report on the Diabetes Distress Scale for Parents of Teens with T1D
Change in autonomy support | Baseline to 9 months
  Participant (young adult) report on the autonomy support sub-scale of the Barriers to Diabetes Adherence Questionnaire
Change in problem solving | Baseline to 9 months
  Participant (young adult) report on the Diabetes Adherence Problem Solving Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Laura Caccavale, PhD, Principal Investigator — Virginia Commonwealth University; Melanie Melanie, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- Children's Hospital of Richmond at Virginia Commonwealth University, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No